CLINICAL TRIAL: NCT03681678
Title: Fractional Carbon Dioxide Laser Therapy of the Vagina for Treatment of Urogenital Symptoms in Women
Brief Title: Laser Therapy for Treatment of Urogenital Symptoms in Women
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Chief Urology, Corewell Health East
Other Study IDs: 2018-142
Record Dates: First submitted 2018-08-03; First posted 2018-09-24 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Genitourinary System; Disorder, Female; Burning Vagina; Dyspareunia; Irritation; Vagina; Menopause Related Conditions; Urinary Incontinence; Urinary Bladder, Overactive; Urinary Tract Infections; Stress Urinary Incontinence
Keywords: Laser Therapy
MeSH Terms: conditions — Dyspareunia; Vaginitis; Urinary Incontinence; Urinary Bladder, Overactive; Urinary Tract Infections; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- fCO2 Laser Therapy Group: Women treated with the fCO2 laser
  Interventions: Device: fCO2 Laser Therapy Group

INTERVENTIONS:
Device: fCO2 Laser Therapy Group — Women enrolled in the study will receive three treatments with the fractional carbon dioxide (fCO2) laser. The interval between treatments is approximately six weeks. Intra-vaginal laser treatments will be delivered at 8 points at each level of the vaginal wall.

SUMMARY:
This is a prospective observational study of women undergoing vaginal treatment with the fractional carbon dioxide (fCO2) laser for various urogenital symptoms.

DETAILED DESCRIPTION:
Fractional carbon dioxide (fCO2) laser treatment of the vaginal tissue has been proposed as a treatment for various genitourinary symptoms, including vaginal itching, burning, dryness, dyspareunia (difficult or painful sexual intercourse), dysuria (painful or difficult urination), nocturia (waking at night to urinate), incontinence (the involuntary loss of urine), urine frequency, urine urgency, and urinary tract infection (UTI).

Case report and case series data suggest that laser treatment of the vaginal tissues is well tolerated by patients and does not pose serious risks to the patient. Several case series demonstrate improvements in vulvovaginal and urinary symptoms, and in sexual function. However, these studies are from a select few centers, are small, and are also biased in that the laser treatment is only available to patients who are able to pay for it. Additionally, most studies report only on vulvovaginal symptoms, despite increasing use of laser for urinary symptoms. Several recent editorials have called for larger studies with longer follow-up and high quality outcome measures. This study has been designed to address these needs.

This is a prospective observational study of women undergoing vaginal treatment with the fCO2 laser for a wide range of patients with vulvovaginal, sexual and/or urologic complaints. The effects of fCO2 therapy will be evaluated by various physical assessments and patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 18 years of age or greater and 90 years of age or less
3. One or more of the following indications for fCO2 laser treatment:

   1. Genitourinary symptoms of menopause, including after natural, medical- induced or surgical menopause
   2. Vaginal dryness, burning, itching or dyspareunia not related to menopause
   3. Stress urinary incontinence
   4. Recurrent urinary tract infections (UTIs), defined as 4 or more in a year
   5. Overactive bladder
4. Must sign the informed consent
5. Must be willing to comply with the study protocol

Exclusion Criteria:

1. Contraindications to fCO2 laser treatment, such as:

   1. Currently implanted synthetic pelvic mesh, sling or tape
   2. Current or previous genital cancers
   3. Radiation to the vaginal or colo-rectal tissue
   4. Currently pregnant or less than 3 months following pregnancy
   5. Undiagnosed vaginal or cervical lesions
2. Patients who have received vaginal fCO2 laser treatment within the past 12 months
3. Patients treated with vaginal estrogen within the past 3 months
4. Patients with undiagnosed vaginal bleeding
5. Active vulvar or vaginal infection, including herpes, candidiasis, etc.
6. Current urinary tract infection (UTI), confirmed by positive urine culture and patient-reported symptoms
7. Pelvic or vaginal surgery with the past 9 months
8. Pelvic organ prolapse beyond the introitus
9. Patient possesses any other characteristics that, per the investigator's judgment, deems them unsuitable (i.e. may increase the patient's risk, may affect the conduct of the study etc.) for the treatment and/or study
10. Participation in an investigational trial that used a study treatment, medication and/or biologic within 6 months or less prior to the date of the screening visit

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women meeting all of the inclusion criteria and non of the exclusion criteria may be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2025-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | fCO2 Laser Therapy Group
Started | 100
Completed | 80 (Primary Endpoint)
Not Completed | 20
Not completed — Lost to Follow-up | 20

BASELINE CHARACTERISTICS:
Arm/Group | fCO2 Laser Therapy Group
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression of Improvement (PGI-I) Score at 4 Weeks After Initial Treatment
Description: PGI-I score is recorded 4 weeks after initial treatment completion. The PGI-I asks the patient to "check the box that best describes how your urinary and/or vaginal symptoms are now, compared with how you symptoms were before you began this study." There are 7 possible responses ranging from 1 to 7, where 1 is "Very Much Better", 2 is "Much Better, 3 is "A Little Bit Better", 4 is "No Change", 5 is "A Little Worse", 6 is "Much Worse", and 7 is "Very Much Worse". A score from 1 to 3 would indicate improvement.
Time Frame: 4 weeks post-initial treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | fCO2 Laser Therapy Group
Number analyzed (Participants) | 80
score on a scale | 2.66 (0.88)

2. Secondary Outcome: Change in Patient Global Impression of Improvement (PGI-I) Score
Description: The average change in patients' PGI-I scores from baseline to 6 months and 36 months post-treatment. The PGI-I asks the patient to "check the one number that best describes how your urinary tract condition is now compared with how it was before your treatment." There are 7 possible responses ranging from 1 to 7, where 1 is "Very Much Better" and 7 is "Very Much Worse". A lower score would represent improvement and a favorable outcome.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

3. Secondary Outcome: Change in Vaginal pH and Overall Vaginal Health on Physical Exam as Measured by the Vaginal Health Inventory Score (VHIS).
Description: The Vaginal Health Inventory Score (VHIS) is an assessment tool, used by providers, to determine if vaginal atrophy is present. Providers perform a vaginal exam and give a score of 1-5 (abnormal to normal, respectively) on each of the following vaginal parameters: elasticity, secretion/fluid volume, vaginal pH, integrity of the epithelium, and lubrication/moisture of the vaginal wall. A VHIS score less than 15 is indicative of vaginal atrophy.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

4. Secondary Outcome: Change in Urinary Symptoms as Measured by the Questionnaire for Urinary Incontinence Diagnosis (QUID).
Description: Patients will complete the QUID, which consists of 6 questions. Responses to the questions indicate the frequency of urinary incontinence. Scores are: 0 (none of the time), 1 (rarely), 2 (once in awhile), 3 (often), 4 (most of the time), or 5 (all of the time). Responses to items 1, 2, and 3 are summed for the Stress Urinary Incontinence Score. Responses to items 4, 5, and 6 are summed for the Urge Incontinence Score.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

5. Secondary Outcome: Change in Overactive Bladder (OAB) Symptoms as Measured by the Overactive Bladder Questionnaire-Short Form (OAB-q SF).
Description: The OAB-q SF consists of two scales assessing symptom bother and health-related quality of life (HR-QOL) in patients with OAB. Each question is rated on a 6 point scale with 1 = Not at all and 6 = A very great deal.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

6. Secondary Outcome: Change in Voiding Diaries.
Description: A 3-day voiding diary will be completed by the patient and evaluated to describe urinary frequency and incontinence episodes.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

7. Secondary Outcome: Change in Sexual Function, Including Dyspareunia Symptoms, as Measured by the Female Sexual Function Inventory (FSFI).
Description: The FSFI consists of 6 subscales related to sexual desire (2 Qs scale 1 worst - 5 best), arousal (4Qs 0 worst - 5 best), lubrication (4Qs 0 worst-5 best), orgasm (3Qs 0 worst - 5 best), satisfaction ( 3Qs 0 worst - 5 best), and pain (3 Qs 0 worst - 5 best). Higher scores indicate higher sexual functioning. Scores range from 2-36. A score of 26.55 has been clinically selected as the cut-off for sexual dysfunction. Scores below this value indicate sexual dysfunction.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

8. Secondary Outcome: Change in Frequency of UTI Occurrences, as Measured by a Positive Urine Culture Test.
Description: A clean catch urine specimen will be collected at each visit. A positive urine dipstick test will have the presence of leukocytes and nitrites accompanied by symptoms (dysuria, bladder pain, and/or urinary frequency).
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

9. Secondary Outcome: Change in Mental Health Status as Measured by the Generalized Anxiety Disorder Questionnaire (GAD-7).
Description: The GAD-7 is a self-reported questionnaire for screening and measuring severity of generalized anxiety disorder. There are 7 questions total, each answer is scored on a scale from 0 = not at all to 3 = nearly every day. Scores greater than or equal to 10 indicate moderate anxiety and further assessment is recommended.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

10. Secondary Outcome: Change in Mental Health Status as Measured by the Patient Health Questionnaire (PHQ-8).
Description: The PHQ-8 is an eight item questionnaire that is a valid diagnostic and severity measure for depressive disorders. Each question is scored from 0 = not at all to 3 = nearly every day. A score of 10 or greater is considered major depression and a score of 20 or more as severe major depression.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

11. Secondary Outcome: Change in Life and Sexual Impact of Vulvovaginal Skin Symptoms.
Description: The Incontinence Quality of Life Questionnaire (I-QOL) is a validated tool to assess the impact of urinary incontinence problems. The I-QOL has 22 incontinent-specific quality of life items all having the following five-point ordinal response scale: 1= Extremely, 2= Quite a Bit, 3= Moderately, 4= A Little, and 5= Not at All. Total I-QOL is a combined score of all items. All 22 items are summed to calculate a total I-QOL score, ranging from 22 to 110, with a high score indicating a better quality of life. The 22 items are broken down into 3 subscales: Avoidance and Limiting Behaviors Score (8 of the 22 items), Psychosocial Impacts Score (9 of the 22 items), and Social Embarrassment Score (5 of the 22 items). Scores are summed based on the same 5-point scale. 1= Extremely, 2= Quite a Bit, 3= Moderately, 4= A Little, and 5= Not at All. A high score indicates a better quality of life.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

12. Secondary Outcome: Change in the Presence of Lactobacillus, Assessed by Vaginal Swab.
Description: Presence or absence of lactobacillus will be collected by the physician via a vaginal swab and assessed under the microscope.
Time Frame: 6 months and 36 months post-initial treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | fCO2 Laser Therapy Group
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 64/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | fCO2 Laser Therapy Group (N=80)
Pudendal nerve pain (Nervous system disorders) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 7 (8)
Urinary Tract Infection (Infections and infestations) | 8 (11)
vaginal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal yeast infection (Infections and infestations) | 4 (4)
Vaginal Burning (Reproductive system and breast disorders) | 2 (3)
Urethral mass (Renal and urinary disorders) | 1 (1)
Bladder pressure (Renal and urinary disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Increase urinary urgency (Renal and urinary disorders) | 4 (4)
Vaginal infection - not specified (Reproductive system and breast disorders) | 1 (1)
ovarian cysts (Reproductive system and breast disorders) | 1 (1)
positive urine dipstick (Renal and urinary disorders) | 1 (2)
Bacterial vaginosis (Infections and infestations) | 5 (6)
Pain during treatment (Injury, poisoning and procedural complications) | 2 (5)
Suspected urinary calculus (Renal and urinary disorders) | 1 (1)
Suspected bacterial vaginosis (Infections and infestations) | 1 (1)
Discomfort with probe insertion (Injury, poisoning and procedural complications) | 4 (4)
Vaginal burning during treatment (Reproductive system and breast disorders) | 5 (5)
Flare of pelvic floor muscle (Musculoskeletal and connective tissue disorders) | 1 (3)
Rash - Allergic reaction to Cipro (Skin and subcutaneous tissue disorders) | 1 (1)
Worsening dyspareunia (Reproductive system and breast disorders) | 1 (1)
Vaginal itching (Reproductive system and breast disorders) | 3 (4)
Vaginal irritation (Reproductive system and breast disorders) | 1 (1)
Numbness to lower extremity and buttock (Nervous system disorders) | 1 (2)
Exacerbation of vaginal atrophy (Reproductive system and breast disorders) | 1 (1)
Left labial itching and redness (Skin and subcutaneous tissue disorders) | 1 (1)
Trauma to introitus during treatment (Injury, poisoning and procedural complications) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03681678/Prot_SAP_000.pdf